CLINICAL TRIAL: NCT07157657
Title: Evaluation of the Efficacy of a Dermal Regeneration Matrix With Photosynthetic Microalgae for the Treatment of Patients With Full-Thickness Skin Wounds: Phase 2 Study
Brief Title: Efficacy of a Photosynthetic Dermal Matrix for the Treatment of Full-Thickness Skin Wounds
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Hospital del Trabajador de Santiago (Other); SymbiOx Inc. (Unknown)
Responsible Party: Principal Investigator, Jose Tomas Egaña, Associate Professor, Pontificia Universidad Catolica de Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEC/21/2024; 24IAT-272741 (Other Grant/Funding Number: CORFO)
Record Dates: First submitted 2025-08-05; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cronic Full-thinkness Skin Wound; Acute Full-thickness Skin Wound
Keywords: Full-thickness skin wounds; Scaffolds for dermal regeneration; Matrix for dermal regeneration; Photosynthetic biomaterials; Oxygen producing biomaterials
MeSH Terms: interventions — GREM1 protein, human

STUDY DESIGN:
Intervention Model Description: This study uses a randomized experimental design. Each enrolled patient will receive both the experimentaland the control treatment. The photosynthetic dermal regeneration matrix (PDRM) will be applied to one wound area, while the standard dermal regeneration matrix (DRM) will be applied to a separate area within the same wound or to a separate, anatomically distinct wound on the same patient. The allocation of wound areas to PDRM or DRM treatment will be randomized to minimize bias and allow within-subject comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with standard or photosynthetic dermal regeneration matrices in same patient. (Experimental): Surgical implantation of dermal regeneration matrices:
  Primary procedure: Participants will receive both a standard dermal regeneration matrix (DRM; control) and a photosynthetic dermal regeneration matrix (PDRM; experimental), which is seeded with Chlamydomonas reinhardtii microalgae. The two matrices will be implanted into randomized areas of the same full-thickness wound or into separate full-thickness wounds on the same patient. A light-emitting dressing will be placed over the wound area to activate photosynthesis in the PDRM, facilitating localized oxygen production.
  Secondary procedure: Approximately 21 days after matrix implantation, once sufficient granulation tissue has formed, an autologous split-thickness skin graft will be applied to the wound areas.
  Interventions: Biological: Surgical implantation with standard (DRM) or photosynthetic dermal regeneration matrices (PDRM) in same patient.; Procedure: Autologous split-thickness skin grafting over implanted matrices

INTERVENTIONS:
Biological: Surgical implantation with standard (DRM) or photosynthetic dermal regeneration matrices (PDRM) in same patient. — Under sterile conditions and appropriate anesthesia, standard dermal regeneration matrices (DRMs) and photosynthetic dermal regeneration matrices (PDRMs), containing live photosynthetic microalgae, are implanted in separate wound areas or in anatomically distinct wounds on the same patient. Each site is then covered with a transparent adhesive dressing. In the experimental (PDRM) area, a light-emitting dressing is applied to stimulate photosynthesis and promote localized oxygen production.
Procedure: Autologous split-thickness skin grafting over implanted matrices — Approximately 21 days after the initial intervention, and once the wound bed meets predefined grafting criteria based on clinical evaluation, an autologous dermo-epidermal skin graft is performed.

SUMMARY:
The goal of this clinical trial is to evaluate whether the incorporation of photosynthetic microalgae into scaffolds for dermal regeneration improves healing outcomes in adult patients with acute and cronic full-thickness skin wounds.

The primary objectives are to determine whether the use of photosynthetic scaffolds enhances wound granulation and reduces infection rates compared to standard dermal regeneration scaffolds. Additionally, the quality of the regenerated skin will be assessed and compared between treatment types.

Participants will:

* Receive treatment with either standard dermal regeneration scaffolds or identical scaffolds containing photosynthetic microalgae. These treatments will be applied either to randomly assigned areas of the same wound or to different wounds on the same patient.
* Undergo regular follow-up assessments to monitor wound healing progress, infection rates, graft integration, and the qualiy of the regenerated skin.
* Complete self-assessment questionnaires regarding their experience and perceived outcomes.

DETAILED DESCRIPTION:
Chronic and acute skin wounds are a significant and growing public health concern, affecting millions of people worldwide and placing a substantial burden on healthcare systems. These wounds, often resulting from underlying conditions such as diabetes, vascular disease, or trauma, can take months or even years to heal, severely impacting patients' quality of life. As global populations age and chronic diseases become more prevalent, the need for more effective wound care solutions is becoming increasingly urgent.

One area of innovation in wound management involves the use of advanced biomaterials that support the body's natural regenerative processes. Dermal regeneration matrices (DRMs) are among the most promising of these technologies, providing a structural scaffold to facilitate tissue repair. However, a major limitation of current DRMs is the poor oxygenation at the wound site during the initial phases of healing-an issue that can delay granulation tissue formation, increase infection risk, and ultimately impair outcomes.

To address this challenge, a novel approach has been developed that incorporates photosynthetic microalgae into the scaffold itself. These microorganisms are capable of producing oxygen when exposed to light, offering a potential means of delivering localized oxygen directly to the wound bed. This photosynthetic dermal regeneration matrix (PDRM) is designed to create a more favorable microenvironment for tissue regeneration by enhancing local oxygen availability in situ.

The present study is a randomized, controlled clinical trial designed to evaluate the safety and efficacy of PDRMs in adult patients with acute and cronic full-thickness skin wounds. Outcomes in wounds treated with PDRMs will be compared to those treated with conventional DRMs. Key endpoints include wound closure, granulation tissue formation, infection rates, graft integration, and overall skin regeneration quality.

If effective, this approach could represent a significant advance in wound care, offering accelerated healing, reduced complications, and improved patient-reported outcomes. The strategy may also broaden the applicability of regenerative therapies in diverse clinical settings by enhancing the functionality of existing biomaterials.

ELIGIBILITY:
Inclusion Criteria:

Patients covered by social insurance law or under the "Complementary Service Sales" (VSC) program, aged 18 years or older.

* Presence of full-thickness skin wounds.
* Wounds with homogeneous granulation tissue.
* Wound size between 25 cm² and 200 cm².
* Signed informed consent to participate in the study.

Exclusion Criteria:

* History of a psychiatric disorder that may impair decision-making or adherence to treatment.
* Presence of an acute medical condition unrelated to the wound at the time of enrollment.
* Wound with exposed bone, tendon, or major blood vessels.
* Psychosocial conditions that may hinder adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Wound granulation rate | From first intervention (Day 0) to readiness of granulation bed for autologus split-thickness sking grafting (up to 21 days).
  Time to wound bed readiness for autologous split-thickness skin grafting, measured in days from the implantation of the dermal regeneration matrix (with or without microalgae) to the clinical determination of over 95% of granulation tissue.
  Wound bed readiness will be assessed using a standardized Clinical Follow-Up Form by at least two independent medical evaluators. Readiness is defined as the presence of well-vascularized, homogeneous granulation tissue deemed suitable for graft acceptance.
  Based on manufacturer data, the expected time to graft readiness in the control (DRM) group is approximately 21 days post-implantation. The microalgae-containing matrix (PDRM) is hypothesized to reduce this time due local oxygen production.

SECONDARY OUTCOMES:
Incidence of wound Infections | From first intervention (Day 0) to readiness of granulation bed for autologus split-thickness sking grafting (up to 21 days).
  The incidence amongst the treated individuals of clinically diagnosed wound infections in areas treated with standard dermal regeneration matrices (DRM) or photosynthetic dermal regeneration matrices (PDRM) will be assessed and compared. Diagnosis will be based on predefined clinical criteria, including signs of erythema, purulent exudate, increased local temperature, and pain, as evaluated by the clinical team.
Patient-Reported Impact | From first intervention (Day 0) to readiness of granulation bed for autologus split-thickness sking grafting (up to 21 days).
  The subjective impact on patients, following treatment with dermal regeneration matrices with or without microalgae (DRM or PDRM) will be assessed using a self-evaluation questionnaire. Five parameters will be assessed (pain, itch, burning, smell, light annoyance), to give a total overall satisfaction percentage related to the presence of the treatment, with percentages closer to 0% indicating less discomfort and more satisfaction.
Autologous graft performance | Following autologous graft implantation (Day 21), patients are monitored periodically for up to 3 months from the date of the original matrix implantation (Day 0).
  The performance of autologous dermo-epidermal grafts placed over control (DRM) or photosynthetic dermal regeneration matrice (PDRM), will be assessed through clinical evaluation. The area of adequate adherence of the autologous dermo-epidermal graft, relative to the initial area of the graft, will be measured. Aditionally, supplementary laboratory tests will be performed, to evaluate the overall health of the patient.
Long-Term Skin Functionality | 3 months after first intervention (Day 0).
  Functional outcomes of the regenerated skin will be assessed through mechanical skin measurements using a Cutometer instrument, to determine and compare the elasticity in areas treated with the different matrices, relative to adjacent healthy skin areas. Skin deformation curves (in mm/sec) will be obtained, and several elasticity parámeter will be calculated and compared between treatments.
Long-Term Skin Appearance | 3 months after first intervention (Day 0).
  Aesthetic outcomes will be evaluated clinically and through patient self-assessment, using the POSAS 3.0 instrument (https://doi.org/10.1007/s11136-022-03244-6), in which an external evaluator, and the patient, score for different perceived characteristics of the treated area, ranging from 1 to 5, with 1 being the best case scenario, and 5 the worst case scenario. Differences betweeen the two treatments will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: José Tomás Egaña, PhD, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital del Trabajador, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
Publication of research articles
Supporting Information: Study Protocol, CSR
Time Frame: Beginning after publication with no end date.

REFERENCES:
- See also: Symbiox website — https://www.symbiox.org/